CLINICAL TRIAL: NCT04972006
Title: Investigating the Acceptability, Feasibility, and Preliminary Efficacy of a Brief, Remote Treatment for Youth Injection Phobia and the Measurement of Cognitive Biases in Youth
Brief Title: Brief, Remote Treatment of Youth Injection Phobia and Measurement of Novel, Disorder-congruent Cognitive Bias Tasks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5992
Record Dates: First submitted 2021-06-16; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Anxiety Disorder of Childhood
Keywords: intensive treatment; remote treatment; cognitive bias; measurement

STUDY DESIGN:
Intervention Model Description: This study uses a multiple baseline design in which participants are assigned to either a one-week, two-week, or three-week baseline period before beginning the study treatment. Participants in all three baseline groups receive the same treatment, both in dose and form.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One week baseline (Experimental): Participants randomized to baseline one will go through a one-week baseline period before beginning the treatment.
  Interventions: Behavioral: Remote, intensive intervention for injection phobia
- Two week baseline (Experimental): Participants randomized to baseline two will go through a two-week baseline period before beginning the treatment.
  Interventions: Behavioral: Remote, intensive intervention for injection phobia
- Three week baseline (Experimental): Participants randomized to baseline three will go through a three-week baseline period before beginning the treatment.
  Interventions: Behavioral: Remote, intensive intervention for injection phobia

INTERVENTIONS:
Behavioral: Remote, intensive intervention for injection phobia — The intervention consists of a 1.5 hour session that provides youth with education about anxiety and a 3 to 4 hour session consisting of graduated exposure to injection fear.

SUMMARY:
This study is investigating the acceptability, feasibility, and preliminary efficacy of a brief, remote treatment for youth injection phobia. It will also be examining the acceptability, feasibility, and initial psychometric properties of three cognitive bias measures adapted or newly developed for youth injection fear.

DETAILED DESCRIPTION:
This study aims to investigate the acceptability, feasibility, and efficacy of a brief, remote treatment for youth injection phobia. There is a pressing need to increase the accessibility, reach, and efficacy of treatments for youth injection fear, as this fear affects approximately 11% of youth and can prevent them from receiving necessary medical procedures or vaccinations. Developing and validating the efficacy of treatments for youth injection fear that are time-efficient, convenient, and broadly accessible will facilitate more widespread targeting of this fear in youth, which could have a meaningful impact on youths' ability to receive medical treatments that involve injections or blood draws. Thus far, separate evidence bases have formed to support the efficacy of brief, intensive treatments for youth specific phobias and other anxiety disorders AND the efficacy of remotely delivered treatments for a range of youth anxiety disorders. However, studies have not yet combined these approaches to investigate their efficacy for treating youth injection phobia. The current study thus serves as the first to specifically examine the clinical utility of using a combined intensive and remote approach to treat youth injection phobia. Investigation into the treatment's impact on youth injection fear will be complemented by information, provided by youths' parents, about the treatment's convenience, acceptability, speed, suitability for the child's specific presentation, and overall helpfulness. Lastly, as a first step towards better understanding the cognitive processing variables that influence the development and maintenance of youth injection fear, the current study will examine the initial acceptability, feasibility, and psychometric properties of adapted or newly developed measures of attentional, interpretation, and memory bias. This study will use a multiple baseline design in which up to 18 youth will be randomly assigned to a one-, two-, or three-week baseline period before beginning the brief, remote intervention. Treatment will consist of two sessions in which the first session provides education about anxiety and lasts approximately 1.5 hours, and the second session consists of gradual exposure to injection-related stimuli and lasts approximately three to four hours. Throughout the study period, youth will complete various measures related to injection fear and related constructs as well as the cognitive bias tasks at three separate time-points.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of specific phobia- blood, injection-injury subtype
* Age between 8 and 16
* Spoken and reading fluency in English
* Third grade reading ability
* Parental availability to participate in treatment study sessions
* Parental spoken and reading fluency in English.

Exclusion Criteria:

* A comorbid, previously assigned diagnosis of attention deficit hyperactivity disorder (ADHD), major depressive disorder (MDD), generalized anxiety disorder (GAD) OR significant parental endorsement of inattentiveness, hyperactivity, prolonged depressed mood, or pervasive generalized worries that are interfering with the child's life at the phone screen level
* A diagnosed learning disorder in reading or information processing
* Parent-reported child unwillingness or lack of ability to participate in cognitive bias tasks (e.g., looking at needle or injection-related imagery, reading basic stories about needles or blood draws)
* Previous and/or concurrent participation in CBT-based, exposure therapy for the fear of injections.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in Fear and Avoidance Ratings | This is a daily measure. Participants will complete it every day for the duration of the study period, which will range between 5 and 7 weeks depending on the participant's baseline assignment.
  Participants will rate their level of fear and avoidance in response to the hypothetical scenario of needing to get a shot. This measure consists of two items, both rated on a scale from 0 (not at all) to 8 (very, very much). The study is interested in looking at the changes in these ratings from the baseline period to the post treatment and two-week follow-up period.

SECONDARY OUTCOMES:
Remote Treatment Acceptability/Feasibility measure | This measure will be administered at the two week follow-up timepoint.
  This measure was adapted for the current study, but is based on the Perceptions of Treatment Questionnaire (Mattis & Ollendick, 1997). The current measure assesses parent's perceptions of the speed, convenience, and helpfulness of the study treatment. The measure consists of 15 items, 11 of which are rated on a Likert scale and 4 of which are free response items. The likert scale items are rated on a 7-point scale, from extremely not (0) to extremely (6).
Measure of the acceptability and feasibility of cognitive bias tasks | This measure will be administered at the two week follow-up timepoint.
  This measure was developed for the purposes of the current study and obtains participants' perspectives about the length, comprehensibility, ease of use, construct validity, and entertainment value of the attentional, interpretation, and memory bias tasks. This measure includes both Likert scale response (9-pt. scale from 0, not at all to 8, very, very much) and free-response items to gain a comprehensive picture of the strengths and limitations of the newly adapted or developed cognitive bias tasks. This measure contains three subscales, each of which corresponds to one of the three cognitive bias tasks (attentional, interpretation, memory). The attentional bias task subscale contains 11 items, the interpretation bias subscale contains 8 items, and the memory bias subscale contains 9 items. The total scale consists of 28 items.
Analysis of test-retest reliability and treatment sensitivity of the attentional bias task | This analysis will include data points from the pre-baseline assessment, the beginning of the first session, and the two week follow-up timepoint.
  Once data collection is complete, it will be possible to analyze the test-retest reliability of the attentional bias task. This will be accomplished by assessing the association between attentional bias indices at pre-treatment and at the beginning of the first session, before treatment has been introduced. Additionally, it will be possible to inspect the treatment sensitivity of the attentional bias task by assessing the difference in magnitude of attentional bias indices before treatment and after treatment at the two-week follow-up time-point.
Analysis of test-retest reliability and treatment sensitivity of the interpretation bias task | This analysis will include data points from the pre-baseline assessment, the beginning of the first session, and the two week follow-up timepoint.
  Once data collection is complete, it will be possible to analyze the test-retest reliability of the interpretation bias task. This will be accomplished by assessing the association between interpretation bias indices at pre-treatment and at the beginning of the first session, before treatment has been introduced. Additionally, it will be possible to inspect the treatment sensitivity of the interpretation bias task by assessing the difference in magnitude of interpretation bias indices before treatment and after treatment at the two-week follow-up time-point.
Analysis of test-retest reliability and treatment sensitivity of the memory bias task | This analysis will include data points from the pre-baseline assessment, the beginning of the first session, and the two week follow-up timepoint.
  Once data collection is complete, it will be possible to analyze the test-retest reliability of the memory bias task. This will be accomplished by assessing the association between the memory bias index at pre-treatment and at the beginning of the first session, before treatment has been introduced. Additionally, it will be possible to inspect the treatment sensitivity of the memory bias task by assessing the difference in magnitude of the memory bias index before treatment and after treatment at the two-week follow-up time-point.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Fenley, MA, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers.